CLINICAL TRIAL: NCT03239210
Title: Effects of Ondansetron in Obsessive-compulsive and Tic Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-01608
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Obsessive-Compulsive Disorder; Tic Disorders; Tourette Syndrome
Keywords: Brain Function; functional magnetic resonance imaging (fMRI); Sensory processing; Obsessive-Compulsive Disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Tic Disorders; Tourette Syndrome | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (OND) (Active Comparator): 24 mg/day for 4 weeks
  Interventions: Drug: Ondansetron
- Placebo (PL) (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — 5-HT3 (serotonin receptor type 3) antagonist commonly used to treat nausea and vomiting
  Other Names: Zofran
  Arms: Ondansetron (OND)
Drug: Placebo — placebo equivalent
  Arms: Placebo (PL)

SUMMARY:
This project investigates the use of 4 weeks of 24 mg/day ondansetron as compared to placebo on symptoms and brain functioning in patients with obsessive-compulsive disorder (OCD) and tic disorders (TD). Patients will be randomized to receive ondansetron or placebo for 4 weeks, with MRI scans and symptom assessments occurring at baseline (before any drug) and at the end of the 4 weeks. Patients will also be asked to come into the lab approximately 2 weeks into the trial for symptom assessments. The investigators hypothesize that after 4 weeks there will be greater reduction from baseline in sensory symptoms and the activation of the insula and sensorimotor cortex compared for ondansetron as compared to placebo.

DETAILED DESCRIPTION:
Many psychiatric disorders are associated with altered sensory experiences arising from within the body. Examples include increased experience of sensations or urges in muscles, skins, joints or visceral organs in Tic/Tourette's Disorders, OCD patients with symptoms of "not just right experiences" or disgust sensitivity, and other disorders such as trichotillomania or excoriation disorder. In OCD, these sensory phenomena occur in approximately half of patients, are associated with earlier age of onset, and may be harder to treat with classic cognitive-behavioral approaches to OCD. Of interest, sensory phenomena in OCD are associated with Tourette's syndrome and respond to pharmacological treatments primarily used for tics. As such, abnormal sensory processing may be a basic mechanism that links various psychiatric disorders.

The process of attending to body sensations is referred to as interoception, abnormality of which may be related to sensory phenomena. Research has revealed a cortical interoceptive circuit involving insula, anterior cingulate cortex (ACC), and sensorimotor cortex. Ondansetron (OND) is a good candidate for the modulation of the above-described interoceptive circuit. It is a selective 5-HT3 (serotonin) receptor antagonist that acts on both peripheral and central receptors. OND has long been used to treat nausea and vomiting due to chemotherapy, radiation therapy, anesthesia, and opioid-induced emesis. It has also been used alone or as adjunctive therapy for the treatment of both OCD and Tourette's disorder, showing some efficacy in small clinical trials. The mechanisms by which ondansetron improves symptoms in OCD and tic disorders are unknown, although the investigator's earlier study found that single doses of ondansetron reduce activation of insula and somatosensory cortex in healthy controls. As a follow-up to this work, the current protocol will compare the effects of 24 mg/day of ondansetron vs. placebo for 4 weeks in patients with OCD or Tic Disorders on symptoms and brain functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be medically healthy, between 18 and 60 years of age
* Fluent (speaking and writing) in English
* Patients must have a current diagnosis of obsessive-compulsive disorder (OCD) or tic disorder (OCD) according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria with moderate or greater disorder severity and moderate or greater severity of sensory phenomena
* Patients must be unmedicated or taking antidepressants, stable for at least 6 weeks

Exclusion Criteria:

* Present or previous diagnosis of any psychosis, bipolar disorder, or major developmental disorder (autism/Asperger's disorder, pervasive developmental disorder). Present diagnosis of alcohol or substance use disorder (moderate or severe) will also be exclusionary.
* Any disability or health problem that prevents them from completing study procedures (e.g. color blindness, severe carpal tunnel syndrome, etc.).
* History of organic mental syndromes, head trauma, migraines, seizures, other central nervous system (CNS) neurological disease, or significant medical illness other than that listed above.
* Pregnant or nursing women will be excluded.
* Subjects with a medical condition or other predisposition that increases the risk of adverse effects when taking ondansetron. These include, but are not limited to, individuals with drug allergies or known hypersensitivity to ondansetron (or other 5-HT3 antagonists), heart disease, congestive heart failure, heart rhythm disorder, congenital long QT syndrome, electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia) or hepatic impairment.
* Subjects who report taking apomorphine will be excluded.
* Subjects with abnormal EKG will either be excluded from participation, or referred to a cardiologist for further assessment of eligibility.
* Subjects with abnormal liver function or electrolytes (as determined by blood test) will be excluded from participation if a study team physician determines it is unsafe for them to participate.
* Cross-reactivity with other 5-HT3 antagonists has been reported, so any individual taking a 5-HT3 antagonist will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Stern, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - The Nathan S. Kline Institute for Psychiatric Research, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Plan The project will be registered and results reported on ClinicalTrials.gov. Neuroimaging data and associated files (e.g. behavioral response data generated during tasks) will be de-identified and provided for use by other researchers. De-identification will include removal of sensitive data from image file headers (e.g. name, date of birth). The anonymized final data set will be made available upon request, with an announcement on the lab website providing information on how to obtain the data. In addition, final data will be uploaded to an appropriate public database, such as the Open fMRI project, for broad availability. Data sharing will comply with local, state, and federal laws and regulations, including the Health Insurance Portability and Accountability Act (HIPAA), as well as institutional policies and review
Time Frame: Data will be made available when the study team has published the outcomes of our primary and secondary analyses.
Access Criteria: A written request must be made to the PI for access to the data. This request will involve providing an abstract detailing the planned analyses and utilization of the data and a signed agreement not to share the data with any other person.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ondansetron (OND) | Placebo (PL)
Started | 33 | 29
Completed | 27 | 24
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by subject (personal reasons) | 2 | 2
Not completed — Withdrawal by subject (reported medical side effects) | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron (OND) | Placebo (PL) | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (9.96) | 29 (12.52) | 30 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 23 | 18 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 21 | 20 | 41
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Activation - Insula Cortex
Description: Change in brain activation is measured by parameter estimate of blood-oxygen-level dependent (BOLD) signal change in the insula cortex. BOLD signal is captured via functional MRI taken during MRI scanning sessions. Participants viewed "body-focused" videos (e.g., close-ups of a brush stroking a hand) alternating with control videos depicting similar types of movements but without body parts (e.g., a pen moving across a table) in an MRI scanner. Analysis examined change in brain activation between baseline and final during the viewing of body-focused videos compared to control videos. The outcome measure is the change in brain activation (Baseline minus Final) averaged across the right and left insula regions of interest.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: Parameter estimate of BOLD Signal Change
Arm/Group | Ondansetron (OND) | Placebo (PL)
Number analyzed (Participants) | 26 | 23
Parameter estimate of BOLD Signal Change | -0.071 (0.21) | -0.0094 (0.23)

2. Primary Outcome: Change in Brain Activation - Somatosensory Cortex
Description: Change in brain activation is measured by parameter estimate of blood-oxygen-level dependent (BOLD) signal change in the somatosensory cortex. BOLD signal is captured via functional MRI taken during MRI scanning sessions. Participants viewed "body-focused" videos (e.g., close-ups of a brush stroking a hand) alternating with control videos depicting similar types of movements but without body parts (e.g., a pen moving across a table) in an MRI scanner. Analysis examined change in brain activation between baseline and final during the viewing of body-focused videos compared to control videos. The outcome measure is the change in brain activation (Baseline minus Final) averaged across the right and left postcentral gyrus regions of interest.
Time Frame: Baseline, Week 4
Measure: Median (95% Confidence Interval); unit: Parameter estimate of BOLD Signal Change
Arm/Group | Ondansetron (OND) | Placebo (PL)
Number analyzed (Participants) | 26 | 23
Parameter estimate of BOLD Signal Change | -0.097 [-0.12 to 0.09] | -0.0052 [-0.14 to 0.08]

3. Secondary Outcome: Change in Sensory Phenomena Scale (SPS) Score
Description: The SPS is a clinician-rated scale that assesses presence or absence of sensory phenomena. It contains a checklist with examples of different types of sensory phenomena, including physical sensations, "just right" sensations, incompleteness, general energy or inner tension buildup, and urges. The total score ranges from 0-15, with higher scores indicating more severe sensory phenomena. A score of 6 or more is defined as moderate or greater severity of sensory phenomena. An decrease in scores indicates severity decreased during the observational period.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ondansetron (OND) | Placebo (PL)
Number analyzed (Participants) | 27 | 24
score on a scale | 1.646 (2.098) | 1.204 (2.143)

4. Secondary Outcome: Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Score
Description: Y-BOCS is designed to rate the severity and type of symptoms in patients with obsessive compulsive disorder. In general, the items depend on the patient's report; however, the final rating is based on the clinical judgement of the interviewer. The scale consists of 10 items summed to determine the level of symptom severity. The total score ranges from 0 to 40 with higher scores indicating greater symptom severity. A decrease in scores indicates symptom severity decreased during the observational period.
Time Frame: Baseline, Week 4
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Ondansetron (OND) | Placebo (PL)
Number analyzed (Participants) | 22 | 22
score on a scale | 2.25 [1.52 to 5.75] | 1 [0.26 to 5.51]

5. Secondary Outcome: Change in Yale Global Tic Severity Scale (YGTSS) Score
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The total score is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity. A decrease in scores indicates severity decreased during the observational period.
Time Frame: Baseline, Week 4
Population: Sample is based on 10 patients with motor/phonic tic symptoms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ondansetron (OND) | Placebo (PL)
Number analyzed (Participants) | 5 | 5
score on a scale | 1.4 (2.97) | 3.6 (6.99)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, as necessary over the period of the trial (typically 4 weeks).
Description: Systematic; Participants filled out the Patient-Rated Inventory of Side Effects (PRISE) at every study visit. The study doctor reviewed each PRISE and monitored AEs throughout the trial.
Arm/Group | Ondansetron (OND) | Placebo (PL)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 22/33 | 12/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron (OND) (N=33) | Placebo (PL) (N=29)
Constipation (Gastrointestinal disorders) | 17 | 1
Headache (Nervous system disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 5 | 1
Dizziness (Nervous system disorders) | 2 | 2
Fatigue (General disorders) | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1
Tremors (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Sleeping too much (Psychiatric disorders) | 1 | 0
Vivid dreams (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Light headed (Nervous system disorders) | 1 | 0
Increase in suicidal ideation (Psychiatric disorders) | 0 | 1
Menstrual irregularity (Reproductive system and breast disorders) | 0 | 1
Frequent urination (Renal and urinary disorders) | 0 | 1
Decreased libido (Psychiatric disorders) | 0 | 1
Transaminitis (transient) (Hepatobiliary disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Poor concentration (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Poor coordination (Nervous system disorders) | 0 | 1
General malaise (General disorders) | 1 | 0
Increased perspiration (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT03239210/Prot_SAP_000.pdf